CLINICAL TRIAL: NCT00778089
Title: Open-Label Study to Evaluate the Immunogenicity of Bovine Collagen in ArteFill® by Skin Testing
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Closed incomplete due to Artes Medical Closing
Sponsor: Suneva Medical, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: D82-3001-07
Record Dates: First submitted 2008-10-21; First posted 2008-10-23 (Estimated); Last update posted 2019-09-27 (Actual); Status verified 2010-03

CONDITIONS: Hypersensitivity
Keywords: skin test; ArteFill; Skin test prior to administration of ArteFill® implant
MeSH Terms: conditions — Hypersensitivity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- Open Label Single Arm (Other): All enrolled subjects will have a skin test composed of Bovine Collagen and Lidocaine.
  Interventions: Device: ArteFill® Skin Test

INTERVENTIONS:
Device: ArteFill® Skin Test — Subjects will receive the ArteFill® Skin Test at Visit 1, Day 0 on the volar forearm. After 30 days, if the test result is negative a second skin test will be administered on the contra volar forearm at Visit, 3, Day 30.

SUMMARY:
The purpose of this study is to assess the clinical utility of the ArteFill® pre-treatment Skin Test in predicting and preventing hypersensitivity reactions to treatment with ArteFill® implant

DETAILED DESCRIPTION:
This is a single-center, open-label study in approximately 485 healthy male and female subjects to obtain 450 evaluable subjects. In this protocol, an ArteFill® Skin Test study will be conducted to evaluate the test's clinical utility to determine the incidence of positive skin reactions to ArteFill®. The results of this skin test study will determine if the risk of a hypersensitivity reaction against ArteFill® without a skin test is no greater than the published historical risk of a hypersensitivity reaction against a Zyderm or Zyplast treatment after a patient demonstrates a negative response to a single Zyderm skin test. Based on prior clinical experience with ArteFill® implant in commercial use outside the United States, it is anticipated that no reactions will be observed. As such, it may be suggested that there is no practical use of the ArteFill® Skin Test for screening patients, and therefore, the test may be eliminated as a requirement prior to treatment with the ArteFill® product as is the clinical practice outside the United States.

ELIGIBILITY:
Inclusion Criteria:

* Subjects 18 years of age or older, male or female.
* Subjects who are healthy and have normal skin on the volar surface of the forearm.
* Subjects willing and able to comply with the requirements of the study.
* Subjects willing and able to comply with the follow-up requirements.
* Subjects willing and able to give written and verbal informed consent.

Exclusion Criteria:

* Subjects who are pregnant, nursing or intend to become pregnant.
* Subjects who have had any form of collagen soft tissue treatment within the last 12 months.
* Subjects who were or are currently being treated with any systemic immunosuppressive therapy including but not limited to chemotherapy agents or corticosteroids (including inhaled or insufflated) within the past 3 months.
* Subjects who were or are currently being treated with any topical OTC drug or prescription therapy on their arms (below the elbow) within the past 3 months.
* Subjects with a history indicative of abnormal immune function (e.g. auto- immune diseases, HIV, cancer, etc).
* Subjects with known lidocaine hypersensitivity.
* Subjects with known sensitivity to bovine collagen.
* Subjects who have a history of dietary beef allergy, undergoing desensitization to beef products or planning to undergo desensitization within the study evaluation period.
* Subjects with severe allergies manifested by a history of anaphylaxis.
* Subject is currently enrolled in an investigational drug or device study.
* Subject has received an investigational drug or an investigational device within 30 days prior to entering this study.
* Subject has any skin pathology or condition that could interfere with the evaluation of the treatment areas.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 498 (Actual)
Dates: Start 2008-07; Primary Completion 2008-12-03 (Actual); Study Completion 2008-12-03 (Actual)

PRIMARY OUTCOMES:
Safety will be assessed by determination of a positive hypersensitivity reaction to the skin test and collection of adverse events. | 60 days

SECONDARY OUTCOMES:
In addition to the primary outcome measure, to assist in assessing the etiology of the reaction, the immune response to the skin test in subjects with positive skin test will be evaluated by measuring serum antibody levels against bovine collagen. | 60 days

CONTACTS AND LOCATIONS:
Overall Officials: David C Wilson, M.D., Principal Investigator — The Education & Research Foundation, Inc.
Locations (1):
- The Education & Research Foundation, Inc., Lynchburg, Virginia, United States